CLINICAL TRIAL: NCT01154764
Title: A Randomized, Open, Crossover Clinical Study to Investigate the Effects of Ketoconazole on the Pharmacokinetics of CG100649 in Healthy Male Volunteers
Brief Title: Trial for Studying Pharmacokinetic Effects of Ketoconazole on CG100649
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CG100649-1-03
Record Dates: First submitted 2010-03-10; First posted 2010-07-01 (Estimated); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: healthy male volunteers
MeSH Terms: interventions — CG100649; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Period 1: CG100649 will be administered alone on Day 1 -After washout period- Period 2: The combination of CG100649 and ketoconazole tabs together on Day 1 followed by ketoconzzole tabs
  Interventions: Drug: CG100649; Drug: Ketoconazole
- Group 2 (Experimental): Period 1: The combination of CG100649 and ketoconazole tabs will be administered together on Day 1, followed by ketoconazole tabs for 4 days, for a total of 5 days.
  -After washout period- Period 2: CG100649 alone
  Interventions: Drug: CG100649; Drug: Ketoconazole

INTERVENTIONS:
Drug: CG100649 — I period: CG 100649 II period: Ketoconalzole + CG100649 at the same time
Drug: Ketoconazole — I period: ketoconazole + CG100649 II period: CG 100649

SUMMARY:
This is a Phase I, open-labeled, randomization and 2x2 Cross trial to compare the pharmacokinetic effects between ketoconazole and CG100649 for healthy male volunteers.

DETAILED DESCRIPTION:
* Adverse Events The whole study discontinuation is determined based on the following criteria with Adverse Events classified using US NCI (National Cancer Institute) 'Common Terminology Criteria for Adverse Events (CTCAE)
* Pharmacokinetic assessment Real sampling times will be used to calculate pharmacokinetic parameters. Concentrations below the lower limit of quantification, samplings which are not applicable, or missing data will be substituted by "<LLOQ", "NA", or "MD" respectively. Pharmacokinetic analyses will be performed on CG100649 only.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-55 years old and weight 50kg above with within 20% of ideal body weight
2. No significant chronic/congenital disease
3. Normal results for lab test
4. Ability of informed consent

Exclusion Criteria:

1. History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
2. History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.
3. History of known hypersensitivity to drugs including CG100649.
4. After taking a rest in sitting position for 3 minutes, subjects who have low blood pressure (Systolic BP ≤ 90 mmHg or Diastolic BP ≤ 50 mmHg) or high blood pressure (Systolic BP ≥ 150 mmHg or Diastolic BP ≥ 100 mmHg).

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, MD, PhD, Principal Investigator — Seoul Asan medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Youn Choi H, Jin SJ, Jung JA, Kim UJ, Ko YJ, Noh YH, Bae KS, Lim HS. Effects of ketoconazole on the pharmacokinetic properties of CG100649, a novel NSAID: a randomized, open-label crossover study in healthy Korean male volunteers. Clin Ther. 2014 Jan 1;36(1):115-25. doi: 10.1016/j.clinthera.2013.12.004. PMID 24417786

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Period 1: CG100649 (1 mg x 6 capsules) once a day, 1 Day Period 2: CG100649 (1 mg x 6 capsules) and ketoconazole tablets (200 mg x 2 tablets) together on Day 1, followed by additional ketoconazole tablets (200 mg x 2 tablets) once a day for 4 days (Days 2-5), for a total of 5 days.
- Group 2: Period 1: CG100649 (1 mg x 6 capsules) and ketoconazole tablets (200 mg x 2 tablets) together on Day 1, followed by additional ketoconazole tablets (200 mg x 2 tablets) once a day for 4 days (Days 2-5), for a total of 5 days.
  Period 2: CG100649 (1 mg x 6 capsules) once a day, 1 Day
Period: Intervention 1 (5days)
Arm/Group | Group 1 | Group 2
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Intervention 2 (5days)
Arm/Group | Group 1 | Group 2
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1 and Group 2: Overall Demographic Character
Arm/Group | Group 1 and Group 2
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Height [Mean (Standard Deviation); unit: centimeters] | 173.2 (4.2)
Weight [Mean (Standard Deviation); unit: kilograms] | 67.0 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 240, 384, and 480 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CG100649 6mg + Ketoconazole 400 mg: CG100649 (1 mg x 6 capsules) and ketoconazole tablets (200 mg x 2 tablets) together on Day 1, followed by additional ketoconazole tablets (200 mg x 2 tablets), once a day for 4 days (Days 2-5), for a total of 5 days.
- CG100649 6mg Single Dosing: CG100649 (1 mg x 6 capsules) once a day single dose
Arm/Group | CG100649 6mg + Ketoconazole 400 mg | CG100649 6mg Single Dosing
Number analyzed (Participants) | 28 | 28
ng/mL | 11.0 (2.4) | 107 (2.4)

2. Primary Outcome: AUClast
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 240, 384, and 480 hours post-dose
Measure: Mean (Standard Deviation); unit: h∙ng/mL
Arm/Group | CG100649 6mg + Ketoconazole 400 mg | CG100649 6mg Single Dosing
Number analyzed (Participants) | 28 | 28
h∙ng/mL | 2685.8 (551.1) | 2074 (442.9)

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Groups:
- CG100649 6mg Single Dosing: CG100649 (1 mg x 6 capsules), once a day
- CG100649+ Ketoconazole: CG100649 (1 mg x 6 capsules) and ketoconazole tablets (200 mg x 2 tablets) together on Day 1, followed by additional ketoconazole tablets (200 mg x 2 tablets), once a day for 4 days (Days 2-5), for a total of 5 days.
Arm/Group | CG100649 6mg Single Dosing | CG100649+ Ketoconazole
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 6/28 | 7/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CG100649 6mg Single Dosing (N=28) | CG100649+ Ketoconazole (N=28)
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Hematuria (Infections and infestations) | 1 | 0
Pyuria (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Clavicle Fractuer (Vascular disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other